CLINICAL TRIAL: NCT06103500
Title: Integrated Clinical Decision Support for Empiric Antibiotic Selection in Sepsis: A Cluster Randomized Cross-Over Trial (IDEAS-CRXO)
Brief Title: Integrated Clinical Decision Support for Empiric Antibiotic Selection in Sepsis
Acronym: IDEAS-CRXO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20230322-01T
Record Dates: First submitted 2023-10-18; First posted 2023-10-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Sepsis; Bacterial Infections; Community-Acquired Infections; Hospital Infection
MeSH Terms: conditions — Sepsis; Bacterial Infections; Community-Acquired Infections; Cross Infection

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Cross-Over Trial
Masking Description: Statistical analyst will be blind to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Decision Support Algorithm for Empiric Antibiotics in Sepsis (Experimental): The planned intervention consists of a pharmacist-facilitated clinical decision support intervention, where pharmacists provide options and recommendations on empiric sepsis antibiotic selection to hospital providers.
  Interventions: Other: Clinical Decision Support Algorithm for Empiric Antibiotics in Sepsis
- Standard of Care (No Intervention): Non-intervention group. No decision support is provided. Patient care is routine.

INTERVENTIONS:
Other: Clinical Decision Support Algorithm for Empiric Antibiotics in Sepsis — A clinical decision support algorithm for empiric antibiotic selection in suspected infection.
  Other Names: Decision Support Tool
  Arms: Clinical Decision Support Algorithm for Empiric Antibiotics in Sepsis

SUMMARY:
As antibiotic resistance increases globally, it becomes more difficult to select empiric antibiotic therapy, particularly in patients with sepsis who stand to benefit from early adequate treatment. In particular it is difficult for clinicians to balance antibiotic stewardship principles (the need to avoid unnecessary prescribing of antibiotics that have an excessively broad spectrum of activity that favour resistance development) and under treatment. The integration of multiple risk variables for resistance are hard for clinicians to translate into clinical action, and is seemingly at odds with the natural inclination to provide heuristic/emotion-based antibiotic selection. The inappropriate treatment of sepsis is not uniformly too broad, or too narrow, and there is a need to optimize and tailor selection of antibiotic therapy to each patient, such that those that are at risk for resistant organisms receive broad therapy, and those that are not at risk, receive narrower antibiotic agents.

Clinicians need support picking the right antibiotic for each patient, and from this they can potentially drive reduction of unnecessarily broad antibiotic prescribing while preserving adequacy of treatment. Individualized clinical prediction models and decision support interventions are promising approaches that meet these needs by improving the classification of patient risk for antibiotic resistant or susceptible infections in sepsis. Unfortunately, few have been validated in the clinical setting and larger rigorous studies are needed to provide the evidence to support broader clinical adoption.

The investigators will perform a cluster randomized cross-over trial of an individualized antibiotic prescribing decision support intervention for providers treating hospitalized patients with suspected sepsis. The aim of this trial is to determine whether a stewardship led clinical decision support intervention can improve antibiotic de-escalation in patients with sepsis while maintaining or improving adequacy of antibiotic coverage. This decision support intervention will be based on a combination of proven decision heuristics (for Gram-positive organisms) and modelled predicted susceptibilities (for Gram-negative organisms) that are individualized to the patient. The primary outcome will be the proportion of patients de-escalated from their initial empiric regimen at 48 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted
2. Age >18 years old
3. Newly started (within 24 hours of assessment for eligibility) on at least one of the following antibiotic(s):

   I. Vancomycin IV II. Linezolid III. Daptomycin IV. Clindamycin V. Cefazolin VI. Cloxacillin VII. Ceftriaxone VIII. Ceftazidime IX. Piperacillin-Tazobactam X. Meropenem (or Imipenem or Ertapenem) XI. Ciprofloxacin
4. Blood cultures ordered (within 12 hours before or after initiation of index antibiotics).

Overall Exclusion:

1. Pregnancy/breastfeeding
2. Documented end-of-life (palliative) care and are/will not be receiving ongoing antibiotic treatment.
3. Already enrolled in the trial.
4. Positive clinical culture results (those with speciation) for the index infection (within 72 hours) already available prior to assessment. Blood cultures with any Gram-positives will be an exclusion. Other cultures that are positive with a Gram-stain result but not speciation will not be an exclusion criteria.
5. Explanatory molecular test (e.g. legionella urinary antigen test, sars-cov-2 testing) within 72 hours prior to assessment.
6. Receipt of antimicrobials (not chronic suppression or prophylaxis) in the prior 24-72 hours (except if started in the outpatient setting or ED prior to admission in the 24-72 hours).
7. The index prescription is a continuation of an antibiotic given for suppressive chronic therapy or long-standing treatment of an established infection.
8. Index antibiotics are peri-operative only or ordered for <24 hours.
9. Cystic fibrosis.
10. Known to be enrolled in a trial that dictates antimicrobial selection.
11. Not eligible for any of the algorithms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of Patients De-escalated | 48 hours
  De-escalation from empiric antibiotic regimen at 48 hours (or at time of discharge if earlier) from receipt of index antibiotics [Binary].

SECONDARY OUTCOMES:
Time to adequate therapy for positive blood cultures | 0-7 days
  Time to adequate therapy for patients with positive blood cultures (hours from time of first index blood culture collection to first dose of agent(s) active against all pathogen(s) in the peri-index positive blood cultures). [Continuous] [Stratified by ampC organisms]
Time to adequate therapy for positive non-screening cultures | 0-7 days
  Time to adequate therapy for patients with positive non-screening cultures including blood cultures (hours from time of first index blood culture collection to first dose of agent(s) active against all pathogen(s) in the peri-index positive cultures). [Continuous][Stratified by ampC organisms]
Number of Patients Receiving Adequate Therapy at 48 hours based on blood cultures | 48 hours
  Receipt of adequate antibiotic therapy within 48 hours (or discharge if earlier) from first index blood culture collection for patients with positive blood cultures (active against all pathogens in peri-index positive blood cultures). [Binary]
Number of Patients Receiving Adequate Therapy at 48 hours based on non-screening cultures | 48 hours
  Receipt of adequate antibiotic therapy within 48 hours (or discharge if earlier) from first index blood culture collection for patients with positive non-screening cultures including blood (active against all pathogens in peri-index positive cultures). [Binary]
Mortality | 90 days
  In-hospital mortality, during index admission, and within 90 days of index event. [Binary]
Length of stay | 0-90 days
  Hospital length of stay on index admission (days) up to 90 days. [Continuous]
De-escalation extent | 48 hours
  Extent of antibiotic de-escalation at 48 hours from index or discharge if earlier (ordinal value up or down the de-escalation cascade, + escalation, - for de-escalation). [Integer from -infinity to infinity]
Antibiotic spectrum at completion | Completion of therapy, up to 90 days
  Antibiotic spectrum rank at 7 days from index antibiotics (or discharge if earlier). [Ordinal]
Number of Patients with C.difficile Infection | 90 days
  Positive stool testing for Clostridioides difficile during index admission, and within 90 days of index. [Binary]
Number of Patients Requiring Dialysis | 90 days
  New requirement for dialysis during index admission, and within 90 days of index. [Binary]
Days of antibiotic therapy | End of index admission, up to 90 days
  Total antibiotic days of therapy (DOT) during the first 7 days from index antibiotics (or prior to discharge if earlier), including by spectrum-level. [Continuous]
Number of Patients with Antibiotic Escalation | 48 hours
  Newly started Gram-positive or Gram-negative coverage, or increases in spectrum of antibiotic therapy, as part of the intervention recommendation. [Binary]
Time to De-escalation | 0-7 days
  Description: Time to antibiotic de-escalation (hours from receipt of index antibiotics). [Continuous][Stratified by ampC organisms]
Number of Patients with Recommended change in Gram-negative coverage | At time of assessment (0 days)
  Recommended change in antibiotic therapy by Gram-negative model. [Binary]
Number of Patients with Accepted change in Gram-negative coverage | Within 24 hours
  Recommended change in antibiotic therapy by Gram-negative model was accepted (acceptance defined as change to some or all of the therapy as recommended within 24 hours of index). [Binary]
Number of Patients with Recommended change in Gram-positive coverage | At time of assessment (0 days)
  Recommended change in antibiotic therapy by Gram-positive algorithm. [Binary]
Number of Patients with Accepted change in Gram-positive coverage | Within 24 hours
  Recommended change in antibiotic therapy by Gram-positive algorithm was accepted and ordered (acceptance defined as change to some or all of the therapy as recommended within 24 hours of index). [Binary]
Number of Patients with Non-recommended escalation at 7 days | 7 days
  Escalation of antibiotic therapy (apart from recommended escalation) within 7 days of receipt of index antibiotics (or prior to discharge if earlier). [Binary]
Number of Patients with ICU admit or mortality | 7 days
  Admitted to ICU on day 7 or not alive at day 7 from receipt of index antibiotics. [Binary]

CONTACTS AND LOCATIONS:
Overall Officials: Derek R Principal Investigator, Principal Investigator — The Ottawa Hospital Research Institute
Locations (3):
- Canada (3):
  - Trillium Health Partners, Mississauga, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario